CLINICAL TRIAL: NCT03423667
Title: Efficacy of N-acetylcysteine on the Craving Symptoms of Abstinent Hospitalized Patients With Cocaine Addiction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruitment (single addictions become rare)
Sponsor: Salvatore Campanella (Other)
Responsible Party: Sponsor-Investigator, Salvatore Campanella, Research Associate FNRS, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUB-Craving NAC
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cocaine Addiction
Keywords: N-acetylcysteine; Craving
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine
- Lactose powder (Placebo Comparator)
  Interventions: Drug: Lactose powder

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine (1200 mg) administered twice a day during 5 days
  Arms: N-acetylcysteine
Drug: Lactose powder — Placebo comparator.
  Arms: Lactose powder

SUMMARY:
Cocaine abuse is associated with serious physical, psychiatric and social problems. Addiction results in the compulsive use of a substance with loss of control and persistence despite the negative consequences.The act of re-engaging in the search for drugs is called relapse and a particularly insidious aspect of addiction is that vulnerability to relapse lasts for many years after stopping drug use.

The main reason why people continue to use cocaine is because of its influence on the reward system.Indeed, this substance makes it possible to increase the level of dopamine, particularly in the nucleus accumbens.This increase in dopamine is not related to the hedonic pleasure that consumption provides. Instead, it imprints a positive value to enhancers and facilitates the learning of reward associations through the modulation of the cortical and subcortical regions of the brain.In other words, it suggests that users become sensitive to a series of stimuli that combine with a rewarding feeling, which drives them to consume when they encounter them.

N-acetylcysteine (NAC) has been used for a long time, mainly as mucolytic. It has also been used as a glutathione antioxidant precursor in the treatment of paracetamol overdose for more than 30 years. NAC has shown beneficial effects in animal models of cocaine addiction by reversing neuroplasticity and reducing the risk of restoring consumer behavior in rodents. Human studies show that NAC is potentially effective in preventing relapse in abstinent patients and ineffective in reducing current consumption.

In this study the investigators will test a sample of newly detoxified (and therefore abstinent) patients who have taken a 3-4 week course of treatment, in order determine if NAC can be a useful medication candidate to avoid relapse in patients with cocaine dependence.

DETAILED DESCRIPTION:
Cocaine abuse is associated with serious physical, psychiatric and social problems. Addiction results in the compulsive use of a substance with loss of control and persistence despite the negative consequences.The act of re-engaging in the search for drugs is called relapse and a particularly insidious aspect of addiction is that vulnerability to relapse lasts for many years after stopping drug use.

The main reason why people continue to use cocaine is because of its influence on the reward system.Indeed, this substance makes it possible to increase the level of dopamine, particularly in the nucleus accumbens.This increase in dopamine is not related to the hedonic pleasure that consumption provides. Instead, it imprints a positive value to enhancers and facilitates the learning of reward associations through the modulation of the cortical and subcortical regions of the brain.In other words, it suggests that users become sensitive to a series of stimuli that combine with a rewarding feeling, which drives them to consume when they encounter them.

Initial investigations regarding the effect of dopamine on the reward system were conducted primarily on the mesolimbic dopaminergic pathway linking the ventral tegmental area to the nucleus accumbens. More recent work has now recognized the role of mesocortical and mesostriatal pathways, but dopamine is far from being the only neurotransmitter involved.

Glutamate also plays a central role in the neuroadaptive changes resulting from chronic exposure to cocaine. Preclinical research has shown that intense exposure to cocaine increases the extracellular level of glutamate in the nucleus accumbens. Cocaine-induced chronic adaptations to glutamatergic homeostasis within the nucleus accumbens include downregulation of the cystine-glutamate (also called xc) exchanger on glial cells and the glial glutamate transporter 1 (GLT-1).

The cystine-glutamate exchanger is an amino acid anti porter that is generally involved in the exchange of extracellular L-cystine (L-Cys2) and intracellular L-glutamate (L-Glu) across the cell plasma membrane. Existing data indicate that these exchanges being diminished, they contribute to abnormal glutamate signaling in the corticostriatal pathway and that these cocaine-induced changes in the Xc system are necessary to restore consumption behavior in the rodent. This imbalance between synaptic and non-synaptic glutamate in the corticostriatal pathway impairs communication between the prefrontal cortex and the nucleus accumbens. As a result, long-term use of cocaine decreases an individual's ability to inhibit the research and consumption behaviors of the product. This results in a relapse syndrome characteristic of addictions.The Xc system would therefore be a potential therapeutic target for the treatment of cocaine addiction.

N-acetylcysteine (NAC) has been used for a long time, mainly as mucolytic. It has also been used as a glutathione antioxidant precursor in the treatment of paracetamol overdose for more than 30 years. NAC has shown beneficial effects in animal models of cocaine addiction by reversing neuroplasticity and reducing the risk of restoring consumer behavior in rodents. One study has even shown that NAC administered to rodents before they consume cocaine prevents the installation of research behavior due to plasticity. Its ability to regulate the activity of the cystine-glutamate antiporter and the biosynthesis of glutathione would be key to its therapeutic efficacy. NAC would also have the ability to reverse the disruption of GLT-1 receptor function. An interesting study has also shown that NAC-treated rats show an attenuation of dopamine increase in the nucleus accumbens when cocaine is taken, which deserves further investigation.

Four studies showed NAC's potential to reduce craving, desire to consume, and cocaine search in abstinent consumers. However these studies present only preliminary data because the samples are not large enough and they are mostly open studies (participants are informed about the nature and dosage of the medication, without placebo group). A more recent study of a larger sample of subjects still actively using cocaine found that NAC reduces craving and increases time to relapse only in a small subset of subjects who are already abstinent, particularly with the highest doses.This study was a double blind study with a placebo group. This suggests that NAC is potentially effective in preventing relapse in abstinent patients and ineffective in reducing current consumption.

A question that arises is the frequency with which NAC should be administered. In the majority of the studies cited above, the product was administered several times over a shorter or longer period. However, studies have shown that a single dose (2400 mg on a human) can have measurable neurochemical effects, although it is not clear that these changes are sufficient to produce measurable changes in behavior.Clinical trials have used doses ranging from 1200 to 3600 mg daily for varying periods of time, and further studies would also be needed to determine the optimal amount to avoid a relapse.

The latest study on the subject suggested that NAC may be useful for preventing relapse of abstinent patients rather than reducing the consumption of patients still taking cocaine. However, this effect was not part of the main assumptions and was highlighted in additional exploratory analyzes. The vast majority of patients in this study were therefore not abstinent.

In this study, therefore, the investigators will only test a sample of newly detoxified (and therefore abstinent) patients who have taken a 3-4 week course of treatment, in order to increase the power of the analyzes and determine if NAC can be a useful medication candidate to avoid relapse in patients with cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Patients addicted to cocaine (according to the DSM V classification)
* Patients admitted for three weeks in the unit 73 of the CHU Brugmann Hospital
* French speaking

Exclusion Criteria:

* Anti-craving or anti-psychotic medication
* Addiction to other drugs (except nicotine or cannabis)
* Neurological medical history
* Psychiatric medical history
* Heavy medical history
* Asthma
* Pregnancy
* Lactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Lickert scale score | Baseline
  Images and videos will be presented to the participants. These will be either neutral or related to drugs consumption (2 images and 1 video of each context). The participants will evaluate their desire to consume, their craving and attraction to each image on a Lickert scale ranging from 0 to 20.
Lickert scale score | 5 days after N-acetylcysteine intake
  Images and videos will be presented to the participants. These will be either neutral or related to drugs consumption (2 images and 1 video of each context). The participants will evaluate their desire to consume, their craving and attraction to each image on a Lickert scale ranging from 0 to 20.
Cocaine craving questionnaire-Brief | Daily from baseline till Day 5 after N-acetylcysteine intake
  The CCQ-Brief consists of 10 items from the CCQ-Now questionnaire, designed to measure a patient's desire to use cocaine. It is intended for use in routine clinical practice (score from 10 till 70)
Relapse rate | 1 month after N-acetylcysteine intake
  Relapse rate
Number of days of abstinence before relapse | From first day of N-acetylcysteine intake until relapse, up to 4 years
  Number of days of abstinence before relapse

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Campanella, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No